CLINICAL TRIAL: NCT04518293
Title: Efficacy and Safety of GMRx2 (a Single Pill Combination Containing Telmisartan/Amlodipine/Indapamide) Compared to Dual Combinations for the Treatment of Hypertension
Brief Title: Efficacy and Safety of GMRx2 Compared to Dual Combinations for the Treatment of Hypertension
Acronym: GMRx2_ACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: George Medicines PTY Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GMRx2-HTN-2020-ACT1
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Amlodipine; Indapamide

STUDY DESIGN:
Intervention Model Description: International, multicenter, randomized, double-blind, active-controlled, parallel group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GMRx2 (Experimental): Telmisartan 20 mg/amlodipine 2.5 mg/indapamide 1.25 mg. At week 6 visit, forced up-titration to telmisartan 40 mg/amlodipine 5 mg/indapamide 2.5 mg
  Interventions: Drug: Telmisartan 20 mg/amlodipine 2.5 mg/indapamide 1.25 mg; Drug: telmisartan 40 mg/amlodipine 5 mg/indapamide 2.5 mg
- Dual - TA (Active Comparator): Telmisartan 20 mg/amlodipine 2.5 mg . At week 6 visit, forced up-titration to telmisartan 40 mg/amlodipine 5 mg
  Interventions: Drug: Telmisartan 20 mg/amlodipine 2.5 mg; Drug: telmisartan 40 mg/amlodipine 5 mg
- Dual - TI (Active Comparator): Telmisartan 20 mg/indapamide 1.25 mg. At week 6 visit, forced up-titration to telmisartan 40 mg/indapamide 2.5 mg
  Interventions: Drug: Telmisartan 20 mg/indapamide 1.25 mg; Drug: telmisartan 40 mg/indapamide 2.5 mg
- Dual - AI (Active Comparator): Amlodipine 2.5 mg/indapamide 1.25 mg. At week 6 visit, forced up-titration to amlodipine 5 mg/indapamide 2.5 mg
  Interventions: Drug: Amlodipine 2.5 mg/indapamide 1.25 mg; Drug: amlodipine 5 mg/indapamide 2.5 mg

INTERVENTIONS:
Drug: Telmisartan 20 mg/amlodipine 2.5 mg/indapamide 1.25 mg — Single pill
  Arms: GMRx2
Drug: telmisartan 40 mg/amlodipine 5 mg/indapamide 2.5 mg — Single pill
  Arms: GMRx2
Drug: Telmisartan 20 mg/amlodipine 2.5 mg — oral tablet
  Arms: Dual - TA
Drug: telmisartan 40 mg/amlodipine 5 mg — oral tablet
  Arms: Dual - TA
Drug: Telmisartan 20 mg/indapamide 1.25 mg — oral tablet
  Arms: Dual - TI
Drug: telmisartan 40 mg/indapamide 2.5 mg — oral tablet
  Arms: Dual - TI
Drug: Amlodipine 2.5 mg/indapamide 1.25 mg — oral tablet
  Arms: Dual - AI
Drug: amlodipine 5 mg/indapamide 2.5 mg — oral tablet
  Arms: Dual - AI

SUMMARY:
Recent hypertension guidelines recommend combination therapy as initial treatment for many or most patients. Several trials suggest triple low-dose combination therapy may be highly effective in terms of achieving blood pressure (BP) control without increasing adverse effects. This trial is designed to investigate the efficacy and safety of GMRx2 in participants with high blood pressure compared to dual combinations.

DETAILED DESCRIPTION:
TRIAL DRUG:

GMRx2: Single pill combinations of telmisartan/amlodipine/indapamide Dose version 2: telmisartan 20mg/amlodipine 2.5mg/indapamide 1.25mg Dose version 3: telmisartan 40mg/amlodipine 5 mg/indapamide 2.5mg INDICATION: Hypertension TRIAL DESIGN: International, multicenter, randomized, double-blind, active controlled, parallel-group.

OBJECTIVES: To investigate the efficacy and safety of GMRx2 compared to dual combinations

INTERVENTION:

Single-Blind Active Run-In Period. Enrolled participants will be asked to discontinue their current BP-lowering drug(s) and undergo a single-blind active run-in period for 4 weeks with GMRx2 dose version 2. Participants will be advised to take the capsule once daily in the morning at approximately the same time each day. For days on which BP is being measured, the capsule should be taken directly after the morning home BP measurement.

Double-Blind Treatment Period. Participants still eligible after the run-in period will be allocated in a double-blind fashion to one of the following 4 randomized groups: GMRx2 dose version 2, or telmisartan 20mg+amlodipine2.5mg, or telmisartan 20mg+indapamide 1.25mg, or amlodipine 2.5mg+indapamide 1.25mg. At week 6 all doses will be doubled.

ELIGIBILITY:
Inclusion Criteria:

At screening visit

1. Provided signed consent to participate in the trial.
2. Adult of age ≥18 years.
3. Attended automated clinic seated mean systolic blood pressure (SBP) (average of last 2 measurements calculated by the device):

140-179 mmHg on 0 BP-lowering drugs, or 130-170 mmHg on 1 BP-lowering drug, or 120-160 mmHg on 2 BP-lowering drugs, or 110-150 mmHg on 3 BP-lowering drugs.

At randomization visit

1. Home seated mean SBP 110-154 mmHg in the week prior to the randomization visit.
2. Adherence of 80-120% to run-in medication.
3. Tolerated run-in medication.
4. Adherence to home BP monitoring schedule: in the week before randomization, at least 6 measures (e.g. ≥2 sets of triplicate measures, ≥3 sets of duplicate measures) including at least 1 morning and 1 evening each with ≥2 measures. Morning is defined as any measure in the am and evening as any measure in the pm. Morning and evening do not have to be same day.

Exclusion Criteria:

At screening visit

1. Receiving 4 or more BP-lowering drugs.
2. Receiving any BP lowering drugs for indications other than hypertension e.g. heart failure
3. Pregnant or had a positive pregnancy test or unwilling to undertake a pregnancy test during the trial and up to 30 days after the discontinuation of the trial medication or breastfeeding or of childbearing age and not using an acceptable method of contraception. Acceptable methods of birth control include hormonal prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method (e.g. condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), or male partner sterilization. Contraception should be used for at least 1 month before the screening visit and until the end of trial participation.
4. Not suitable for participation in a clinical trial according to local ethical or regulatory requirements related to severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2).
5. Contraindication, including hypersensitivity (e.g. anaphylaxis or angioedema), to the active run-in treatment or to any of the trial medication options in the four randomized groups.
6. Current/history of transient ischemic attack, stroke, or hypertensive encephalopathy.
7. Current/history of acute coronary syndrome, unstable angina, myocardial infarction, percutaneous transluminal coronary revascularization, or coronary artery bypass graft.
8. Current atrial fibrillation. Patients with a history of paroxysmal atrial fibrillation are potentially eligible as long as there has been no episode in the last 3 months, while patient with a history of persistent or permanent atrial fibrillation are not eligible.
9. Current/history of New York Heart Association class III and IV congestive heart failure.
10. Current/history of a known secondary cause of hypertension, such as primary aldosteronism, renal artery stenosis, pheochromocytoma, or Cushing's syndrome.
11. Current/history of substantially uncontrolled diabetes (HbA1c > 11.0%) within last three months.
12. Current/history of end-stage renal disease or anuria or estimated glomerular filtration rate (eGFR) <60 ml/min/1.73m2.
13. Electrolyte levels that would be regarded as contraindications for any of the potential treatment arms e.g. serum sodium <132mmol/l or >148mmol/l serum potassium <3.1 mmol/l or >5.6 mmol/l.
14. Current/history of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 times the upper limit of normal range within 6 months.
15. Current concomitant illness or physical impairment or mental condition that in the judgment of the investigator could interfere with the effective conduct of the trial or constitutes a significant risk to the participants' well-being.
16. Arm circumference that is too large (>55 cm) or too small (<15-24 cm) to allow accurate measurement of BP.
17. Currently taking or might need during the trial, a concomitant treatment which is known to interact with one or more of the trial medications: digoxin, lithium, diabetics receiving aliskiren, moderate and strong CYP3A4 inhibitors (e.g. ritonavir, ketoconazole, diltiazem], simvastatin >20 mg/day, immunosuppressants.
18. Might need treatment with drugs that are prohibited during the trial: other antihypertensive drugs, endothelin receptor antagonists, neprilysin inhibitors, or other drugs that may affect BP.
19. Current surgical or medical condition that might significantly alter the absorption, distribution, metabolism, or excretion of trial drugs such as prior major gastrointestinal tract surgery (e.g. gastrectomy, lap band, or bowel resection) or acute flare of inflammatory bowel disease within one year.
20. Individuals working >2 nightshifts per week.
21. Participated in any investigative drug or device trial within the previous 30 days.
22. History of alcohol or drug abuse within 12 months.

At randomization visit

1. Unable to adhere to the trial procedures during the run-in treatment period.
2. Any of the following which in the investigator's judgment may compromise the safety of the participant if randomized to the trial medications:

   1. High or low clinic BP levels even in the light of the values for home BP that are available for that participant. The exact levels of BP are not specified, since there is clinical uncertainty as to the relevance of BP levels which are high or low in clinic only; for example, the clinical relevance of 'whitecoat hypertension' is uncertain.
   2. High or low home diastolic BP (DBP) levels. The exact levels of DBP is not specified, reflecting clinical uncertainty of the implications of isolated diastolic hypertension. However, home DBP values of >99 mmHg may typically be considered as requiring treatment intensification, and such participants would not be suitable for randomization.
   3. Any abnormal laboratory value which in the judgment of the investigator could interfere with the effective conduct of the trial or constitutes a significant risk to the participants' well-being.
   4. Fulfilling any of the exclusion criteria mentioned for the screening visit, when verified again at randomization visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1385 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Rodgers, Professor, Principal Investigator — The George Institute
Locations (86):
- United States (30):
  - Elite Clinical Studies, Phoenix, Arizona
  - Headlands Research, Scottsdale, Arizona
  - Quality of Life Medical & Research Associates, Tucson, Arizona
  - Valiance Clinical Research, South Gate, California
  - Valiance Clinical Research, Tarzana, California
  - Clinical Research of Brandon, Brandon, Florida
  - Inpatient Research Clinic, Hialeah, Florida
  - Multi-Speciality Research Associates, Lake City, Florida
  - Suncoast Research Group, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Ocala Research Institute, Ocala, Florida
  - Suncoast Research Associates, St. Petersburg, Florida
  - Accel Research, St. Petersburg, Florida
  - Precision Research Center, Tampa, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Buckhead Primary Care Research, Snellville, Georgia
  - Loyola University, Maywood, Illinois
  - Meridian Clinical Research, Baton Rouge, Louisiana
  - Meridian Clinical Research, Endwell, New York
  - Javarra Research, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - The University of Tennessee Health Science Center, Memphis, Tennessee
  - ACRC Trials - Southwest Medical Village, Austin, Texas
  - ACRC Trials - Premier Family Physicians, Austin, Texas
  - ACRC Trials - Family Medicine Associates of Texas, Carlton, Texas
  - Synergy Groups Medical, Houston, Texas
  - Synergy Groups Medical, Missouri City, Texas
  - North Hills Medical Research, North Richland Hills, Texas
  - ACRC Trials - Village Health Partners, Plano, Texas
  - Meridian Clinical Research, Portsmouth, Virginia
- Australia (6):
  - Castle Hill Medical Centre, Castle Hill, New South Wales
  - Princess Alexandra Hospital - Hypertension Unit, Brisbane, Queensland
  - Hudson Institute of Medical Research, Clayton, Victoria
  - Barwon Health, Geelong University Hospital, Geelong, Victoria
  - Curtin University, Bentley, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Czechia (3):
  - Private Cardiologic Ambulance, Medicus Services s.r.o, Brandýs nad Labem, Central Bohemia
  - EDUMED, s.r.o, Broumov, Kralovehradsky
  - EDUMED, s.r.o, Jaroměř, Kralovehradsky
- New Zealand (2):
  - Middlemore Clinical Trials, Otahuhu, Auckland
  - Gisborne Hospital, Gisborne
- Poland (10):
  - Medical University of Gdansk, Gdansk, Gdansk
  - Futuremeds, Wroclaw, Wroclaw
  - Medical University of Gdansk, Gdansk
  - Pratia Katowice Medical Centre, Katowice
  - Nowodworskie Medical Center, Nowy Dwór Mazowiecki
  - Medical Center Pratia Poznan, Poznan
  - ETG Network, Skierniewice
  - The Medical University of Warsaw, Warsaw
  - EMC Instytut Medyczny S.A, Wroclaw
  - Futuremeds, Wroclaw
- Sri Lanka (10):
  - Clinical Medicine Academic & Research Centre, Colombo
  - Institute of Cardiology, National Hospital of Sri Lanka, Colombo
  - Colombo South Teaching Hospital, Dehiwala
  - Karapitiya Teaching Hospital, Galle
  - Jafna Teaching Hospital, Jaffna
  - Kandy National Hospital, Kandy
  - Kurunegala Teaching Hospital, Kurunegala
  - Negombo District General Hospital, Negombo
  - Sri Jayawardenapura General Hospital, Nugegoda
  - Colombo North Teaching Hospital, Ragama
- United Kingdom (25):
  - Steploe Medical Centre, Soham, Cambridgeshire
  - Ashfields Primary Care Centre, Sandbach, Cheshire
  - Newquay Medical, Newquay, Cornwall
  - Royal Primary care Ashgate, Chesterfield, Derbyshire
  - Carmel Medical Practice, Darlington, Durham
  - PRC Leciester, Leicester, East Midlands
  - Portmill Surgery, Hitchin, Herts.
  - Layton Medical Centre, Blackpool, Lancashire
  - Waterloo Medical Centre, Blackpool, Lancashire
  - Burbage Surgery, Hinckley, Leicestershire
  - Belmont Health Centre, Harrow, London
  - The Adam Practice, Upton, Poole
  - Heart of bath Medical Partnership, Bath, Somerset
  - West Walk Surgery, Bristol, Somerset
  - Tyntesfield Medical Group, Nailsea, Somerset
  - Clifton Medical centre, Rotherham, South Yorkshire
  - Ely Bridge, Cardiff, Wales
  - Atherstone Surgery, Atherstone, Warwickshire
  - Lakeside Surgery, Coventry, West Midlands
  - Sherbourne Medical Centre, Royal Leamington Spa, West Midlands
  - Hathaway Surgery, Chippenham, Wiltshire
  - Rowden Surgery, Chippenham, Wiltshire
  - Trowbridge Health Centre, Trowbridge, Wiltshire
  - Bart's NHS Trust, London
  - Ecclesfield group Practice, Sheffield

IPD SHARING:
Plan to Share IPD: No
If the sponsor receives a request for study data, then such requests will be reviewed by sponsor following completion of regulatory submissions and review, and with support from members of the GMRX2 steering committee who will advise on the scientific merit and integrity of the proposed analysis.

REFERENCES:
- [Derived] Rodgers A, Salam A, Schutte AE, Cushman WC, de Silva HA, Di Tanna GL, Grobbee DE, Narkiewicz K, Ojji DB, Poulter NR, Schlaich MP, Oparil S, Spiering W, Williams B, Wright JT Jr, Lakshman P, Uluwattage W, Hay P, Pereira T, Amarasena N, Ranasinghe G, Gianacas C, Shanthakumar M, Liu X, Wang N, Gnanenthiran SR, Whelton PK; GMRx2 Investigators. Efficacy and safety of a novel low-dose triple single-pill combination of telmisartan, amlodipine and indapamide, compared with dual combinations for treatment of hypertension: a randomised, double-blind, active-controlled, international clinical trial. Lancet. 2024 Oct 19;404(10462):1536-1546. doi: 10.1016/S0140-6736(24)01744-6. PMID 39426836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 83 study centers across 7 countries (Australia [6], Czech Republic [2], Great Britain [25], New Zealand [2], Poland [9], Sri Lanka [14], and USA [25]).
Groups:
- Dual - TA: Telmisartan 20 mg/amlodipine 2.5 mg . At week 6 visit, forced up-titration to telmisartan 40 mg/amlodipine 5 mg
  Telmisartan 20 mg/amlodipine 2.5 mg .: oral tablet
  telmisartan 40 mg/amlodipine 5 mg: oral tablet
Period: Single, Active run-in (4 Weeks)
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Started | 2244 (A total of 2,244 screened participants entered in the GMRx2 run-in treatment period, during which participants were all switched from existing regimens to GMRx2 Dose 2.) | 0 | 0 | 0
Completed (Enrolled participants completed single-blind active run-in period on GMRx2 and were subsequently randomized to blinded treatment arms.) | 1385 (Following run-in, 1385 participants were randomized with a 2:1:1:1 ratio of GMRx2: Dual-TA: Dual-TI: Dual-AI during the double-blind period.) | 0 | 0 | 0
Not Completed | 859 | 0 | 0 | 0
Period: Double-blind
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Started (Enrolled patients completed screening and unblinded active run-in on GMRx2, and were subsequently randomised to a blinded treatment arm.) | 551 | 282 | 276 | 276
Completed (Completion of trial is defined as attending Week 12/Visit Follow-Up 2 and Week 16/Visit End of Trial.) | 527 | 273 | 259 | 259
Not Completed | 24 | 9 | 17 | 17

BASELINE CHARACTERISTICS:
Groups:
- Dual - TA: Telmisartan 20 mg/amlodipine 2.5 mg. At week 6 visit, forced up-titration to telmisartan 40 mg/amlodipine 5 mg
  Telmisartan 20 mg/amlodipine 2.5 mg: oral tablet
  telmisartan 40 mg/amlodipine 5 mg: oral tablet
- Total: Total of all reporting groups
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI | Total
Number analyzed (Participants) | 551 | 282 | 276 | 276 | 1385
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.1 (11.28) | 58.7 (11.41) | 59.2 (10.29) | 58.9 (11.32) | 59.0 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 276 | 145 | 143 | 148 | 712
  Male | 275 | 137 | 133 | 128 | 673
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 31 | 30 | 35 | 159
  Not Hispanic or Latino | 487 | 250 | 246 | 241 | 1224
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 272 | 135 | 132 | 134 | 673
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 3 | 1 | 9
  Black or African American | 30 | 11 | 13 | 16 | 70
  White | 246 | 132 | 128 | 125 | 631
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 8 | 4 | 4 | 4 | 20
  United States | 83 | 44 | 42 | 49 | 218
  Sri Lanka | 260 | 131 | 128 | 127 | 646
  Czechia | 4 | 2 | 3 | 2 | 11
  Poland | 4 | 2 | 2 | 1 | 9
  United Kingdom | 138 | 73 | 72 | 68 | 351
  Australia | 54 | 26 | 25 | 25 | 130
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — Population: Data on BMI was reported for 545, 281 and 273 participants for GMRx2, dual-TA and dual-TI groups.
  Kg/m^2
    number analyzed (Participants) | 545 | 281 | 273 | 276 | 1375
    (all) | 28.87 (5.688) | 28.68 (5.735) | 29.05 (5.686) | 28.82 (6.022) | 28.86 (5.761)
Weight [Mean (Standard Deviation); unit: Kg] — Population: Data on weight was reported for 545, 281 and 273 participants for GMRx2, dual-TA and dual-TI groups.
  Kg
    number analyzed (Participants) | 545 | 281 | 273 | 276 | 1375
    (all) | 79.09 (20.714) | 78.19 (19.995) | 79.38 (20.623) | 78.03 (20.859) | 78.75 (20.565)
Height [Mean (Standard Deviation); unit: cm] — Population: Data on height was reported for 545, 281 and 273 participants for GMRx2, dual-TA and dual-TI groups.
  cm
    number analyzed (Participants) | 545 | 281 | 273 | 276 | 1375
    (all) | 164.72 (11.054) | 164.47 (10.659) | 164.54 (11.566) | 163.84 (11.702) | 164.46 (11.204)
Smoking [Count of Participants; unit: Participants]
  Never | 431 | 207 | 198 | 211 | 1047
  Ex-smoker | 92 | 60 | 64 | 50 | 266
  Current smoker | 28 | 15 | 14 | 15 | 72
Alcohol [Count of Participants; unit: Participants]
  Currently drink alcohol once a week or more | 179 | 101 | 96 | 105 | 481
  Not currently drinking | 372 | 181 | 180 | 171 | 904
Pre-Screening 12-Lead ECG [Count of Participants; unit: Participants]
  Normal | 402 | 214 | 215 | 210 | 1041
  Atrial fibrillation | 0 | 0 | 0 | 0 | 0
  Any other abnormalities | 120 | 57 | 48 | 52 | 277
  Missing | 29 | 11 | 13 | 14 | 67
Hypertension Status at Screening [Count of Participants; unit: Participants]
  Office BP<140/90 mmHg | 197 | 92 | 96 | 104 | 489
  Office BP≥140/90 mmHg | 354 | 190 | 180 | 172 | 896
Number of Prior BP Treatments at Screening [Count of Participants; unit: Participants]
  0 | 65 | 27 | 28 | 24 | 144
  1 | 193 | 110 | 83 | 87 | 473
  2 | 217 | 105 | 112 | 121 | 555
  3 | 76 | 40 | 53 | 44 | 213

OUTCOME MEASURES:

1. Primary Outcome: Difference in Change in Home Seated Mean Systolic Blood Pressure (SBP) From Randomization to Week 12
Description: The primary outcome measure is difference in change in average home SBP for GMRx2 vs each dual combination evaluated from randomization to Week 12. The change in home SBP from randomization for all treatment arms was measured using least squares (LS) mean change. The pairwise comparisons between GMRx2 and dual treatments in change in home SBP were estimated using LS means difference and are described in the statistical analysis.
Time Frame: Week 12
Population: Analysis was performed on all participants who had been randomized. Participants were analyzed in the treatment group to which they had been randomized.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
mmHg | -4.0 (0.45) | 1.4 (0.60) | -1.5 (0.51) | 0.4 (0.62)
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The LS means (LSM) difference (95% CI) in home seated SBP reduction was calculated between GMRx2 and dual-TA arms; Test type: Other — The difference between GMRx2 and dual-TA at Week 12 was estimated using a mixed model for repeated measures (MMRM); p < .0001, MIANALYZE procedure; LS Means Difference = -5.44, 95% CI 2-sided [-6.774 to -4.107], Standard Error of Mean 0.680
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The LSM difference (95% CI) in home SBP reduction was calculated between GMRx2 and dual-TI arms; Test type: Other — The difference between GMRx2 and dual-TI at Week 12 was estimated using a MMRM; p < .0001, MIANALYZE procedure; LS Means Difference = -2.49, 95% CI 2-sided [-3.723 to -1.251], Standard Error of Mean 0.630
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The LSM difference (95% CI) in home SBP reduction was calculated between GMRx2 and dual-AI arms; Test type: Other — The difference between GMRx2 and dual-AI at Week 12 was estimated using a MMRM; p < .0001, MIANALYZE procedure; LS Means Difference = -4.42, 95% CI 2-sided [-5.758 to -3.091], Standard Error of Mean 0.680

2. Secondary Outcome: Difference in Change in Clinic Seated Mean Systolic Blood Pressure (SBP) From Randomization to Week 12
Description: Difference in change in average clinic SBP for GMRx2 vs each dual combination was evaluated from randomization to Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
mmHg | -5.5 (0.55) | 0.1 (0.85) | -1.2 (1.02) | 0.9 (0.86)
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The LSM difference (95% CI) in clinic SBP reduction was calculated between GMRx2 between dual-TA arms; Test type: Other — The difference between GMRx2 and dual-TA at Week 12 was estimated using a MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -5.60, 95% CI 2-sided [-7.307 to -3.902], Standard Error of Mean 0.863
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The LSM difference (95% CI) in clinic SBP reduction was calculated between GMRx2 and dual-TI arms; Test type: Other — The difference between GMRx2 and dual-TI at Week 12 was estimated using a MMRM; p = 0.0005, Mixed Models Analysis; LS Means Difference = -4.33, 95% CI 2-sided [-6.718 to -1.933], Standard Error of Mean 1.212
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The LSM difference (95% CI) in clinic SBP reduction was calculated between GMRx2 and dual-AI arms; Test type: Other — The difference between GMRx2 and dual-AI at Week 12 was estimated using a MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -6.33, 95% CI 2-sided [-7.984 to -4.680], Standard Error of Mean 0.837

3. Secondary Outcome: Difference in Change in Clinic Seated Mean Systolic Blood Pressure (SBP) From Randomization to Week 6
Description: Difference in change in average clinic SBP for GMRx2 vs each dual combination was evaluated from randomization to Week 6.
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
mmHg | -0.8 (0.50) | 4.2 (0.88) | 2.7 (0.96) | 4.5 (1.02)
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The LSM difference (95% CI) in clinic SBP reduction was calculated between GMRx2 and dual-TA arms; Test type: Other — The difference between GMRx2 and dual-TA at Week 6 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -5.01, 95% CI 2-sided [-6.703 to -3.317], Standard Error of Mean 0.858
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The LSM difference (95% CI) in clinic SBP reduction was calculated between GMRx2 and dual-TI arms; Test type: Other — The difference between GMRx2 and dual-TI at Week 6 was estimated using MMRM; p = 0.0002, Mixed Models Analysis; LS Means Difference = -3.50, 95% CI 2-sided [-5.293 to -1.700], Standard Error of Mean 0.910
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The LSM difference (95% CI) in clinic SBP reduction was calculated between GMRx2 and dual-AI arms; Test type: Other — The difference between GMRx2 and dual-AI at Week 6 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -5.35, 95% CI 2-sided [-7.251 to -3.444], Standard Error of Mean 0.965

4. Secondary Outcome: Difference in Change in Clinic Seated Mean Diastolic Blood Pressure (DBP) From Randomization to Week 12
Description: Difference in change in average clinic DBP for GMRx2 vs each dual combination was evaluated from randomization to Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
mmHg | -3.4 (0.42) | 0.4 (0.52) | 0.2 (0.56) | 1.1 (0.61)
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The LSM difference (95% CI) in clinic DBP reduction was calculated between GMRx2 and dual-TA arms; Test type: Other — The difference between GMRx2 and dual-TA at Week 12 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -3.72, 95% CI 2-sided [-4.692 to -2.757], Standard Error of Mean 0.490
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The LSM difference (95% CI) in clinic DBP reduction was calculated between GMRx2 and dual-TI arms; Test type: Other — The difference between GMRx2 and dual-TI at Week 12 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -3.51, 95% CI 2-sided [-4.897 to -2.128], Standard Error of Mean 0.702
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The LSM difference (95% CI) in clinic DBP reduction was calculated between GMRx2 and dual-AI arms; Test type: Other — The difference between GMRx2 and dual-AI at Week 12 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -4.50, 95% CI 2-sided [-5.812 to -3.189], Standard Error of Mean 0.665

5. Secondary Outcome: Difference in Change in Clinic Seated Mean Diastolic Blood Pressure (DBP) From Randomization to Week 6
Description: Difference in change in average clinic DBP for GMRx2 vs each dual combination was evaluated from randomization to Week 6.
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
mmHg | -0.7 (0.38) | 1.7 (0.57) | 1.6 (0.57) | 3.1 (0.57)
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The LSM difference (95% CI) in clinic DBP reduction was calculated between GMRx2 and dual-TA arms; Test type: Other — The difference between GMRx2 and dual-TA at Week 6 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -2.43, 95% CI 2-sided [-3.392 to -1.469], Standard Error of Mean 0.487
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The LSM difference (95% CI) in clinic DBP reduction was calculated between GMRx2 and dual-TI arms; Test type: Other — The difference between GMRx2 and dual-TI at Week 6 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -2.29, 95% CI 2-sided [-3.371 to -1.201], Standard Error of Mean 0.550
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The LSM difference (95% CI) in clinic DBP reduction was calculated between GMRx2 and dual-AI arms; Test type: Other — The difference between GMRx2 and dual-AI at Week 6 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -3.77, 95% CI 2-sided [-4.882 to -2.664], Standard Error of Mean 0.562

6. Secondary Outcome: Percentage of Participants With Clinic Seated Mean Systolic Blood Pressure (SBP) <140 and Diastolic Blood Pressure (DBP) <90 mmHg at Week 12
Description: The percentage of participants achieving averaged clinic SBP <140 mmHg and DBP <90 mmHg at Week 12 was evaluated.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 407 | 173 | 167 | 146
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The difference between GMRx2 and TA at Week 12 was estimated using Generalized Estimating Equation; Test type: Other; p = 0.0003, Wald test; Risk Difference (RD) = 12.52, 95% CI 2-sided [5.630 to 19.487]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The difference between GMRx2 and TI at Week 12 was estimated using Generalized Estimating Equation; Test type: Other; p = 0.0001, Wald test; Risk Difference (RD) = 13.36, 95% CI 2-sided [6.392 to 20.394]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The difference between GMRx2 and AI at Week 12 was estimated using Generalized Estimating Equation; Test type: Other; p < .0001, Wald test; Risk Difference (RD) = 20.97, 95% CI 2-sided [13.812 to 28.013]

7. Secondary Outcome: Percentage of Participants With Clinic Seated Mean Systolic Blood Pressure (SBP) <140 and Diastolic Blood Pressure (DBP) <90 mmHg at Week 6
Description: The percentage of participants achieving averaged clinic SBP <140 mmHg and DBP <80 mmHg at Week 6 was evaluated.
Time Frame: Week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 346 | 148 | 151 | 122
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The difference between GMRx2 and TA at Week 6 was estimated using Generalized Estimating Equation; Test type: Other; p = 0.0044, Wald test; Risk Difference (RD) = 10.31, 95% CI 2-sided [3.044 to 17.535]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The difference between GMRx2 and TI at Week 6 was estimated using Generalized Estimating Equation; Test type: Other; p = 0.0262, Wald test; Risk Difference (RD) = 8.08, 95% CI 2-sided [0.804 to 15.373]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The difference between GMRx2 and AI at Week 6 was estimated using Generalized Estimating Equation; Test type: Other; p < .0001, Wald test; Risk Difference (RD) = 18.59, 95% CI 2-sided [11.201 to 25.746]

8. Secondary Outcome: Percentage of Participants With Clinic Seated Mean Systolic Blood Pressure (SBP) <130 and Diastolic Blood Pressure (DBP) <80 mmHg at Week 12
Description: The percentage of participants achieving averaged clinic SBP <130 mmHg and DBP <80 mmHg at Week 12 was evaluated.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 218 | 65 | 76 | 59
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The difference between GMRx2 and TA at Week 12 was estimated using Generalized Estimating Equation; Test type: Other; p < .0001, Wald test; Risk Difference (RD) = 16.51, 95% CI 2-sided [9.707 to 22.837]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The difference between GMRx2 and TI at Week 12 was estimated using Generalized Estimating Equation; Test type: Other; p = 0.0004, Wald test; Risk Difference (RD) = 12.03, 95% CI 2-sided [4.982 to 18.658]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The difference between GMRx2 and AI at Week 12 was estimated using Generalized Estimating Equation; Test type: Other; p < .0001, Wald test; Risk Difference (RD) = 18.19, 95% CI 2-sided [11.412 to 24.432]

9. Secondary Outcome: Percentage of Participants With Clinic Seated Mean Systolic Blood Pressure (SBP) <130 and Diastolic Blood Pressure (DBP) <80 mmHg at Week 6
Description: The percentage of participants achieving averaged clinic SBP <130 mmHg and DBP <80 mmHg at Week 6 was evaluated.
Time Frame: Week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 167 | 56 | 59 | 50
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The difference between GMRx2 and TA at Week 6 was estimated using Generalized Estimating Equation; Test type: Other; p = 0.0007, Wald test; Risk Difference (RD) = 10.45, 95% CI 2-sided [3.993 to 16.433]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The difference between GMRx2 and TI at Week 6 was estimated using Generalized Estimating Equation; Test type: Other; p = 0.0046, Wald test; Risk Difference (RD) = 8.93, 95% CI 2-sided [2.337 to 15.058]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; Test type: Other; p < .0001, Wald test; Risk Difference (RD) = 12.19, 95% CI 2-sided [5.792 to 18.073]

10. Secondary Outcome: Difference in Change in Home Seated Mean Systolic Blood Pressure (SBP) From Randomization to Week 6
Description: Difference in change in average home SBP for GMRx2 vs each dual combination was evaluated from randomization to Week 6.
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
mmHg | -0.9 (0.40) | 5.2 (0.57) | 2.1 (0.49) | 4.2 (0.56)
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The LSM difference (95% CI) in home SBP reduction was calculated between GMRx2 and dual-TA arms; Test type: Other — The difference between GMRx2 and dual-TA at Week 6 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -6.11, 95% CI 2-sided [-7.086 to -5.144], Standard Error of Mean 0.495
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The LSM difference (95% CI) in home SBP reduction was calculated between GMRx2 and dual-TI arms; Test type: Other — The difference between GMRx2 and dual-TI at Week 6 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -3.00, 95% CI 2-sided [-4.060 to -1.932], Standard Error of Mean 0.543
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The LSM difference (95% CI) in home SBP reduction was calculated between GMRx2 and dual-AI arms; Test type: Other — The difference between GMRx2 and dual-AI at Week 6 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -5.09, 95% CI 2-sided [-6.274 to -3.912], Standard Error of Mean 0.603

11. Secondary Outcome: Difference in Change in Home Seated Mean Diastolic Blood Pressure (DBP) From Randomization to Week 12
Description: Difference in change in average home DBP for GMRx2 vs each dual combination was evaluated from randomization to Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
mmHg | -2.9 (0.28) | 0.5 (0.32) | -0.8 (0.35) | 0.7 (0.45)
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The LSM difference (95% CI) in home DBP reduction was calculated between GMRx2 and dual-TA arms; Test type: Other — The difference between GMRx2 and dual-TA at Week 12 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -3.35, 95% CI 2-sided [-4.069 to -2.632], Standard Error of Mean 0.364
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The LSM difference (95% CI) in home DBP reduction was calculated between GMRx2 and dual-TI arms; Test type: Other — The difference between GMRx2 and dual-TI at Week 12 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -2.10, 95% CI 2-sided [-2.998 to -1.200], Standard Error of Mean 0.456
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The LSM difference (95% CI) in home DBP reduction was calculated between GMRx2 and dual-AI arms; Test type: Other — The difference between GMRx2 and dual-AI at Week 12 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -3.63, 95% CI 2-sided [-4.617 to -2.649], Standard Error of Mean 0.499

12. Secondary Outcome: Difference in Change in Home Seated Mean Diastolic Blood Pressure (DBP) From Randomization to Week 6
Description: Difference in change in average home DBP for GMRx2 vs each dual combination was evaluated from randomization to Week 6.
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
mmHg | -0.7 (0.29) | 2.5 (0.39) | 1.3 (0.40) | 2.5 (0.41)
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The LSM difference (95% CI) in home DBP reduction was calculated between GMRx2 and dual-TA arms; Test type: Other — The difference between GMRx2 and dual-TA at Week 6 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -3.52, 95% CI 2-sided [-4.137 to -2.908], Standard Error of Mean 0.311
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The LSM difference (95% CI) in home DBP reduction was calculated between GMRx2 and dual-TI arms; Test type: Other — The difference between GMRx2 and dual-TI at Week 6 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -2.09, 95% CI 2-sided [-2.803 to -1.376], Standard Error of Mean 0.361
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The LSM difference (95% CI) in home DBP reduction was calculated between GMRx2 and dual-AI arms; Test type: Other — The difference between GMRx2 and dual-AI at Week 6 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -3.58, 95% CI 2-sided [-4.446 to -2.713], Standard Error of Mean 0.439

13. Secondary Outcome: Difference in Change in Trough Home Seated Mean Systolic Blood Pressure (SBP) From Randomization to Week 12
Description: Difference in change in trough home SBP for GMRx2 vs each dual combination was evaluated from randomization to Week 12. Trough values were measured before morning dose of the study medication.
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
mmHg | -4.0 (0.48) | 1.6 (0.59) | -2.1 (0.58) | -0.2 (0.63)
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The LSM difference (95% CI) in trough (i.e. before morning dose) home SBP reduction was calculated between GMRx2 and dual-TA arms; Test type: Other — The difference between GMRx2 and dual-TA at Week 12 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -5.58, 95% CI 2-sided [-6.983 to -4.169], Standard Error of Mean 0.713
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The LSM difference (95% CI) in trough (i.e. before morning dose) home SBP reduction was calculated between GMRx2 and dual-TI arms; Test type: Other — The difference between GMRx2 and dual-TI at Week 12 was estimated using MMRM; p = 0.0043, Mixed Models Analysis; LS Means Difference = -1.91, 95% CI 2-sided [-3.218 to -0.607], Standard Error of Mean 0.662
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The LSM difference (95% CI) in trough (i.e. before morning dose) home SBP reduction was calculated between GMRx2 and dual-AI arms; Test type: Other — The difference between GMRx2 and dual-AI at Week 12 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -3.74, 95% CI 2-sided [-5.214 to -2.274], Standard Error of Mean 0.745

14. Secondary Outcome: Difference in Change in Trough Home Seated Mean Systolic Blood Pressure (SBP) From Randomization to Week 6
Description: Difference in change in trough home SBP for GMRx2 vs each dual combination was evaluated from randomization to Week 6. Trough values were measured before morning dose of the study medication.
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
mmHg | -0.9 (0.41) | 5.3 (0.66) | 1.8 (0.61) | 3.5 (0.57)
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; [analysis description as in outcome 13, analysis 1]; Test type: Other — The difference between GMRx2 and dual-TA at Week 6 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -6.25, 95% CI 2-sided [-7.324 to -5.168], Standard Error of Mean 0.546
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; [analysis description as in outcome 13, analysis 2]; Test type: Other — The difference between GMRx2 and dual-TI at Week 6 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -2.72, 95% CI 2-sided [-3.941 to -1.507], Standard Error of Mean 0.616
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; [analysis description as in outcome 13, analysis 3]; Test type: Other — The difference between GMRx2 and dual-AI at Week 6 was estimated using MMRM; p < .0001, Mixed Models Analysis; LS Means Difference = -4.43, 95% CI 2-sided [-5.489 to -3.368], Standard Error of Mean 0.537

15. Secondary Outcome: Percentage of Participants With Home Seated Mean Systolic Blood Pressure (SBP) <135 and Diastolic Blood Pressure (DBP) <85 mmHg at Week 12
Description: The percentage of participants achieving averaged home SBP <135 mmHg and DBP <85 mmHg at week 12 was calculated.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 398 | 162 | 176 | 155
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The difference between GMRx2 and TA at Week 12 was estimated using Generalized Estimating Equation; Test type: Other; p < .0001, Wald test; Risk Difference (RD) = 14.79, 95% CI 2-sided [7.749 to 21.824]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The difference between GMRx2 and TI at Week 12 was estimated using Generalized Estimating Equation; Test type: Other; p = 0.0146, Wald test; Risk Difference (RD) = 8.46, 95% CI 2-sided [1.580 to 15.501]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The difference between GMRx2 and AI at Week 12 was estimated using Generalized Estimating Equation; Test type: Other; p < .0001, Wald test; Risk Difference (RD) = 16.07, 95% CI 2-sided [8.953 to 23.171]

16. Secondary Outcome: Percentage of Participants With Home Seated Mean Systolic Blood Pressure (SBP) <135 and Diastolic Blood Pressure (DBP) <85 mmHg at Week 6
Description: The percentage of participants achieving averaged home SBP <135 mmHg and DBP <85 mmHg at Week 6 was evaluated.
Time Frame: Week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 346 | 126 | 155 | 123
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The difference between GMRx2 and TA at Week 6 was estimated using Generalized Estimating Equation; Test type: Other; p < .0001, Wald test; Risk Difference (RD) = 18.11, 95% CI 2-sided [10.778 to 25.226]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The difference between GMRx2 and TI at Week 12 was estimated using Generalized Estimating Equation; Test type: Other; p = 0.0674, Wald test; Risk Difference (RD) = 6.64, 95% CI 2-sided [-0.613 to 13.926]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The difference between GMRx2 and AI at Week 12 was estimated using Generalized Estimating Equation; Test type: Other; p < .0001, Wald test; Risk Difference (RD) = 18.23, 95% CI 2-sided [10.839 to 25.392]

17. Secondary Outcome: Percentage of Participants With Home Seated Mean Systolic Blood Pressure (SBP) <130 and Diastolic Blood Pressure (DBP) <80 mmHg at Week 12
Description: The percentage of participants achieving averaged home SBP <130 mmHg and DBP <80 mmHg at Week 12 was evaluated.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 308 | 109 | 121 | 91
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The difference between GMRx2 and TA at Week 12 was estimated using Generalized Estimating Equation; Test type: Other; p < .0001, Wald test; Risk Difference (RD) = 17.25, 95% CI 2-sided [9.902 to 24.286]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The difference between GMRx2 and TI at Week 12 was estimated using Generalized Estimating Equation; Test type: Other; p = 0.0010, Wald test; Risk Difference (RD) = 12.06, 95% CI 2-sided [4.632 to 19.293]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The difference between GMRx2 and AI at Week 12 was estimated using Generalized Estimating Equation; Test type: Other; p < .0001, Wald test; Risk Difference (RD) = 22.93, 95% CI 2-sided [15.622 to 29.796]

18. Secondary Outcome: Percentage of Participants With Home Seated Mean Systolic Blood Pressure (SBP) <130 and Diastolic Blood Pressure (DBP) <80 mmHg at Week 6
Description: The percentage of participants achieving averaged home SBP <130 mmHg and DBP <80 mmHg at Week 6 was evaluated.
Time Frame: Week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 247 | 74 | 90 | 79
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The difference between GMRx2 and TA at Week 6 was estimated using Generalized Estimating Equation; Test type: Other; p < .0001, Wald test; Risk Difference (RD) = 18.59, 95% CI 2-sided [11.579 to 25.124]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The difference between GMRx2 and TI at Week 6 was estimated using Generalized Estimating Equation; Test type: Other; p = 0.0005, Wald test; Risk Difference (RD) = 12.22, 95% CI 2-sided [4.963 to 19.123]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The difference between GMRx2 and AI at Week 6 was estimated using Generalized Estimating Equation; Test type: Other; p < .0001, Wald test; Risk Difference (RD) = 16.20, 95% CI 2-sided [9.060 to 22.914]

19. Other Pre Specified Outcome: Percentage of Participants Discontinued Trial Medication Due to Adverse Event (AE)/Serious Adverse Event (SAE) From Randomization to Week 12
Description: The primary safety outcome is the proportion of participants who discontinued trial medication due to an AE or SAE from randomization to follow-up at Week 12.
Time Frame: Week 12
Population: Analysis was done on the safety set which included all participants who had taken at least one dose of study treatment, including during Period 1 single-blind run-in. For the analysis of the safety outcomes, participants were analyzed in the treatment group that was received.
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 11 | 3 | 4 | 4
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants discontinuing trial medication due to AE/SAE at Week 12 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 0.93, 95% CI 2-sided [-1.529 to 2.768]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants discontinuing trial medication due to AE/SAE at Week 12 was calculated between GMRx2 and dual-TI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 0.55, 95% CI 2-sided [-2.098 to 2.475]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants discontinuing trial medication due to AE/SAE at Week 12 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 0.55, 95% CI 2-sided [-2.098 to 2.475]

20. Other Pre Specified Outcome: Percentage of Participants Discontinued Trial Medication Due to Adverse Event (AE)/Serious Adverse Event (SAE) From Randomization to Week 6
Description: The secondary safety outcome is the proportion of participants who discontinued trial medication due to AE/SAE from randomization to follow-up at Week 6.
Time Frame: Week 6
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 5 | 3 | 1 | 3

21. Other Pre Specified Outcome: Percentage of Participants With a Serious Adverse Event (SAE) From Randomization to Week 12
Description: The secondary safety outcome is the proportion of participants with at least one SAE from randomization to follow-up at Week 12.
Time Frame: At Week 12
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 17 | 6 | 7 | 6

22. Other Pre Specified Outcome: Percentage of Participants With Serious Adverse Event (SAE) From Randomization to Week 6
Description: The secondary safety outcome is the proportion of participants with at least one SAE from randomization to follow-up at Week 6.
Time Frame: Week 6
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 12 | 4 | 4 | 6

23. Other Pre Specified Outcome: Percentage of Participants With Symptomatic Hypotension From Randomization to Week 12
Description: The secondary safety outcome is the proportion of participants who experienced at least one symptomatic hypotension episode from randomization to follow-up at Week 12.
Time Frame: Week 12
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 32 | 5 | 11 | 4

24. Other Pre Specified Outcome: Percentage of Participants With Symptomatic Hypotension From Randomization to Week 6
Description: The secondary safety outcome is the proportion of participants who experienced at least one symptomatic hypotension episode from randomization to follow-up at Week 6.
Time Frame: Week 6
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 15 | 3 | 1 | 2

25. Other Pre Specified Outcome: Percentage of Participants With Serum Sodium Concentration Below 135 mmol/l at Week 12
Description: The secondary safety outcome is the proportion of participants with serum sodium <135 mmol/L at follow-up Week 12.
Time Frame: Week 12
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 40 | 9 | 19 | 10
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with serum sodium concentration below 135 mmol/l at Week 12 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 4.07, 95% CI 2-sided [0.494 to 7.116]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with serum sodium concentration below 135 mmol/l at Week 12 was calculated between GMRx2 and dual-TI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 0.38, 95% CI 2-sided [-3.927 to 4.020]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants with serum sodium concentration below 135 mmol/l at Week 12 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 3.64, 95% CI 2-sided [-0.070 to 6.764]

26. Other Pre Specified Outcome: Percentage of Participants With Serum Sodium Concentration Below 135 mmol/l at Week 6
Description: The secondary safety outcome is the proportion of participants with serum sodium <135 mmol/L at follow-up Week 6.
Time Frame: Week 6
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 26 | 6 | 8 | 11
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with serum sodium concentration below 135 mmol/l at Week 6 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 2.59, 95% CI 2-sided [-0.500 to 5.136]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with serum sodium concentration below 135 mmol/l at Week 6 was calculated between GMRx2 and dual-TI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 1.82, 95% CI 2-sided [-1.513 to 4.517]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants with serum sodium concentration below 135 mmol/l at Week 6 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 0.73, 95% CI 2-sided [-2.855 to 3.633]

27. Other Pre Specified Outcome: Percentage of Participants With Serum Sodium Concentration Above 145 mmol/l at Week 12
Description: The secondary safety outcome is the proportion of participants with serum sodium >145 mmol/L at follow-up Week 12.
Time Frame: Week 12
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 29 | 15 | 16 | 13
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with serum sodium concentration above 145 mmol/l at Week 12 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = -0.06, 95% CI 2-sided [-3.911 to 3.129]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with serum sodium concentration above 145 mmol/l at Week 12 was calculated between GMRx2 and dual-TI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = -0.53, 95% CI 2-sided [-4.519 to 2.744]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants with serum sodium concentration above 145 mmol/l at Week 12 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 0.55, 95% CI 2-sided [-3.228 to 3.647]

28. Other Pre Specified Outcome: Percentage of Participants With Serum Sodium Concentration Above 145 mmol/l at Week 6
Description: The secondary safety outcome is the proportion of participants with serum sodium >145 mmol/L at follow-up Week 6.
Time Frame: Week 6
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 26 | 14 | 8 | 15
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with serum sodium concentration above 145 mmol/l at Week 6 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = -0.25, 95% CI 2-sided [-3.993 to 2.816]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with serum sodium concentration above 145 mmol/l at Week 6 was calculated between GMRx2 and dual-TI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 1.82, 95% CI 2-sided [-1.513 to 4.517]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; [analysis description as in outcome 28, analysis 2]; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = -0.72, 95% CI 2-sided [-4.596 to 2.440]

29. Other Pre Specified Outcome: Percentage of Participants With Serum Potassium Concentration Below 3.5 mmol/l at Week 12
Description: The secondary safety outcome is the proportion of participants with serum potassium concentration <3.5 mmol/L at follow-up Week 12.
Time Frame: Week 12
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 37 | 0 | 13 | 35
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with serum potassium concentration below 3.5 mmol/l at Week 12 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 6.72, 95% CI 2-sided [4.196 to 9.222]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with serum potassium concentration below 3.5 mmol/l at Week 12 was calculated between GMRx2 and dual-TI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 2.00, 95% CI 2-sided [-1.883 to 5.257]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants with serum potassium concentration below 3.5 mmol/l at Week 12 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = -5.97, 95% CI 2-sided [-10.979 to -1.600]

30. Other Pre Specified Outcome: Percentage of Participants With Serum Potassium Concentration Below 3.5 mmol/l at Week 6
Description: The secondary safety outcome is the proportion of participants with serum potassium concentration below 3.5 mmol/l at follow-up Week 6.
Time Frame: Week 6
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 27 | 5 | 10 | 21
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with serum potassium concentration below 3.5 mmol/l at Week 6 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 3.13, 95% CI 2-sided [0.123 to 5.632]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with serum potassium concentration below 3.5 mmol/l at Week 6 was calculated between GMRx2 and dual-TI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 1.28, 95% CI 2-sided [-2.245 to 4.134]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants with serum potassium concentration below 3.5 mmol/l at Week 6 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = -2.71, 95% CI 2-sided [-6.968 to 0.819]

31. Other Pre Specified Outcome: Percentage of Participants With Serum Potassium Concentration Above 5.5 mmol/l at Week 12
Description: The secondary safety outcome is proportion of participants with serum potassium concentration >5.5 mmol/l at follow-up Week 12.
Time Frame: Week 12
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 5 | 0 | 0 | 1
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with serum potassium concentration above 5.5 mmol/l at Week 12 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 0.91, 95% CI 2-sided [-0.863 to 2.231]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with serum potassium concentration above 5.5 mmol/l at Week 12 was calculated between GMRx2 and dual-TI arms; Test type: Other; Risk Difference (RD) = 0.91, 95% CI 2-sided [-0.897 to 2.231]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants with serum potassium concentration above 5.5 mmol/l at Week 12 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 0.55, 95% CI 2-sided [-1.494 to 1.913]

32. Other Pre Specified Outcome: Percentage of Participants With Serum Potassium Concentration Above 5.5 mmol/l at Week 6
Description: The secondary safety outcome is proportion of participants with serum potassium concentration >5.5 mmol/L at follow-up Week 6.
Time Frame: Week 6
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 2 | 1 | 1 | 0
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with serum potassium concentration above 5.5 mmol/l at Week 6 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 0.01, 95% CI 2-sided [-1.931 to 1.149]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with serum potassium concentration above 5.5 mmol/l at Week 6 was calculated between GMRx2 and dual-TI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 0.00, 95% CI 2-sided [-1.979 to 1.143]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants with serum potassium concentration above 5.5 mmol/l at Week 6 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 0.36, 95% CI 2-sided [-1.374 to 1.453]

33. Other Pre Specified Outcome: Percentage of Participants With Estimated Glomerular Filtration Rate (eGFR) Drop of Over 30% From Randomization to Week 12
Description: The secondary safety outcome was the proportion of participants with an eGFR drop of over 30% from randomization to follow-up at Week 12.
Time Frame: Week 12
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 8 | 3 | 1 | 1
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with eGFR drop of over 30% at Week 12 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 0.39, 95% CI 2-sided [-2.014 to 2.087]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with eGFR drop of over 30% at Week 12 was calculated between GMRx2 and dual-TI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 1.09, 95% CI 2-sided [-1.015 to 2.633]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants with eGFR drop of over 30% at Week 12 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 1.09, 95% CI 2-sided [-1.015 to 2.633]

34. Other Pre Specified Outcome: Percentage of Participants With Estimated Glomerular Filtration Rate (eGFR) Drop of Over 30% From Randomization to Week 6
Description: The secondary safety outcome is the proportion of participants with an eGFR drop of over 30% from randomization to follow-up at Week 6.
Time Frame: Week 6
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 5 | 3 | 4 | 3
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with eGFR drop of over 30% at Week 6 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = -0.16, 95% CI 2-sided [-2.501 to 1.385]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with eGFR drop of over 30% at Week 6 was calculated between GMRx2 and dual-TI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = -0.54, 95% CI 2-sided [-3.078 to 1.108]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants with eGFR drop of over 30% at Week 6 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = -0.18, 95% CI 2-sided [-2.571 to 1.370]

35. Other Pre Specified Outcome: Percentage of Participants With Serum Sodium <135mmol/L or >145 mmol/L, and/or Serum Potassium <3.5 mmol/L or >5.5mmol/L at Follow-up Week 12
Description: The secondary safety outcome is the proportion of participants with serum sodium <135mmol/L or >145 mmol/L, and/or serum potassium <3.5 mmol/L or >5.5mmol/L at follow-up Week 12.
Time Frame: Week 12
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 105 | 24 | 44 | 57
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with serum sodium <135mmol/L or >145 mmol/L, and/or serum potassium <3.5 mmol/L or >5.5mmol/L at Week 12 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 10.55, 95% CI 2-sided [5.422 to 15.138]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with serum sodium <135mmol/L or >145 mmol/L, and/or serum potassium <3.5 mmol/L or >5.5mmol/L at Week 12 was calculated between GMRx2 and dual-TI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 3.11, 95% CI 2-sided [-2.776 to 8.490]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants with serum sodium <135mmol/L or >145 mmol/L, and/or serum potassium <3.5 mmol/L or >5.5mmol/L at Week 12 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = -1.60, 95% CI 2-sided [-7.807 to 4.174]

36. Other Pre Specified Outcome: Percentage of Participants With Serum Sodium <135 mmol/L or >145 mmol/L, and/or Serum Potassium <3.5 mmol/L or >5.5 mmol/L at Week 6
Description: The secondary safety outcome is proportion of participants with serum sodium <135 mmol/L or >145 mmol/L, and/or serum potassium <3.5 mmol/L or >5.5 mmol/L at follow-up Week 6.
Time Frame: Week 6
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 79 | 25 | 26 | 44
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with serum sodium <135mmol/L or >145 mmol/L, and/or serum potassium <3.5 mmol/L or >5.5mmol/L at Week 6 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 5.47, 95% CI 2-sided [0.531 to 9.867]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with serum sodium <135mmol/L or >145 mmol/L, and/or serum potassium <3.5 mmol/L or >5.5mmol/L at Week 6 was calculated between GMRx2 and dual-TI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = 4.92, 95% CI 2-sided [-0.136 to 9.397]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants with serum sodium <135mmol/L or >145 mmol/L, and/or serum potassium <3.5 mmol/L or >5.5mmol/L at Week 6 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; Risk Difference (RD) = -1.60, 95% CI 2-sided [-7.299 to 3.567]

37. Other Pre Specified Outcome: Percentage of Participants With Orthostatic Hypotension at Week 6
Description: The secondary safety outcome is the proportion of participants with orthostatic hypotension at follow-up Week 6.
Time Frame: Week 6
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 27 | 14 | 20 | 15
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with orthostatic hypotension at Week 6 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; p = 0.9677, Wald test; Risk Difference (RD) = -0.06, 95% CI 2-sided [-3.825 to 3.019]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with orthostatic hypotension at Week 6 was calculated between GMRx2 and dual-TI arms; Test type: Other; p = 0.1952, Wald test; Risk Difference (RD) = -2.35, 95% CI 2-sided [-6.550 to 1.125]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants with orthostatic hypotension at Week 6 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; p = 0.7453, Wald test; Risk Difference (RD) = -0.53, 95% CI 2-sided [-4.428 to 2.642]

38. Other Pre Specified Outcome: Percentage of Participants With Orthostatic Hypotension at Week 12
Description: The secondary safety outcome is the proportion of participants with orthostatic hypotension at follow-up Week 12.
Time Frame: Week 12
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 28 | 14 | 21 | 20
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with orthostatic hypotension at Week 12 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; p = 0.9415, Wald test; Risk Difference (RD) = 0.12, 95% CI 2-sided [-3.657 to 3.222]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with orthostatic hypotension at Week 12 was calculated between GMRx2 and dual-TI arms; Test type: Other; p = 0.1719, Wald test; Risk Difference (RD) = -2.53, 95% CI 2-sided [-6.799 to 1.019]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants with orthostatic hypotension at Week 12 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; p = 0.2342, Wald test; Risk Difference (RD) = -2.16, 95% CI 2-sided [-6.380 to 1.326]

39. Other Pre Specified Outcome: Percentage of Participants With Orthostatic Hypertension at Week 6
Description: The secondary safety outcome is the proportion of participants with orthostatic hypertension at follow-up Week 6.
Time Frame: Week 6
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 119 | 69 | 57 | 66
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with orthostatic hypertension at Week 6 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; p = 0.3548, Wald test; Risk Difference (RD) = -2.87, 95% CI 2-sided [-9.316 to 3.215]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with orthostatic hypertension at Week 6 was calculated between GMRx2 and dual-TI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; p = 0.7529, Wald test; Risk Difference (RD) = 0.94, 95% CI 2-sided [-5.356 to 6.800]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants with orthostatic hypertension at Week 6 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; p = 0.4563, Wald test; Risk Difference (RD) = -2.32, 95% CI 2-sided [-8.791 to 3.772]

40. Other Pre Specified Outcome: Percentage of Participants With Orthostatic Hypertension at Week 12
Description: The secondary safety outcome is the proportion of participants with orthostatic hypertension at follow-up Week 12.
Time Frame: Week 12
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GMRx2 | Dual - TA | Dual - TI | Dual - AI
Number analyzed (Participants) | 551 | 282 | 276 | 276
Participants | 112 | 57 | 66 | 57
Statistical Analysis 1: Comparison: GMRx2 vs Dual - TA; The Risk difference (95% CI) in percentage of participants with orthostatic hypertension at Week 12 was calculated between GMRx2 and dual-TA arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; p = 0.9691, Wald test; Risk Difference (RD) = 0.11, 95% CI 2-sided [-6.063 to 5.859]
Statistical Analysis 2: Comparison: GMRx2 vs Dual - TI; The Risk difference (95% CI) in percentage of participants with orthostatic hypertension at Week 12 was calculated between GMRx2 and dual-TI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; p = 0.2454, Wald test; Risk Difference (RD) = -3.59, 95% CI 2-sided [-10.018 to 2.462]
Statistical Analysis 3: Comparison: GMRx2 vs Dual - AI; The Risk difference (95% CI) in percentage of participants with orthostatic hypertension at Week 12 was calculated between GMRx2 and dual-AI arms; Test type: Other — 95% CI for risk difference utilized Newcombe estimation method; p = 0.9130, Wald test; Risk Difference (RD) = -0.33, 95% CI 2-sided [-6.583 to 5.488]

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: The safety set included all participants who had taken at least one dose of study treatment, including during Period 1 single-blind run-in. For the analysis of the safety outcomes, participants were analyzed in the treatment group that was received during the double-blind treatment period. Safety analysis was also performed for the participants who were not randomized to any of the treatment groups.
Groups:
- Not Randomized: Participants who were run-in failure and were not randomized (most common reason being home seated mean SBP of 120-154 mmHg in week prior to randomization visit and other reason).
Arm/Group | Not Randomized | GMRx2 | Dual - TA | Dual - TI | Dual - AI
All-Cause Mortality (participants affected / at risk) | 0/859 | 0/551 | 0/282 | 0/276 | 0/276
Serious Adverse Events (participants affected / at risk) | 15/859 | 22/551 | 11/282 | 14/276 | 8/276
Other Adverse Events (participants affected / at risk) | 136/859 | 306/551 | 139/282 | 142/276 | 136/276
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Not Randomized (N=859) | GMRx2 (N=551) | Dual - TA (N=282) | Dual - TI (N=276) | Dual - AI (N=276)
COVID-19 (Infections and infestations) | 9 | 14 | 6 | 12 | 7
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Retroperitoneal fibrosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Lacrimal gland abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 2 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Not Randomized (N=859) | GMRx2 (N=551) | Dual - TA (N=282) | Dual - TI (N=276) | Dual - AI (N=276)
Blood glucose increased (Investigations) | 0 | 42 | 15 | 19 | 26
Blood uric acid increased (Investigations) | 0 | 37 | 9 | 19 | 23
Glomerular filtration rate decreased (Investigations) | 10 | 20 | 9 | 15 | 14
Blood sodium decreased (Investigations) | 0 | 24 | 10 | 12 | 10
Hyponatremia (Metabolism and nutrition disorders) | 19 | 28 | 12 | 14 | 16
Hypokalemia (Metabolism and nutrition disorders) | 10 | 28 | 6 | 8 | 20
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 15 | 13 | 9 | 8
Headache (Nervous system disorders) | 14 | 30 | 10 | 13 | 9
Blood cholesterol increased (Investigations) | 0 | 22 | 17 | 9 | 4
Blood creatinine increased (Investigations) | 0 | 28 | 8 | 12 | 4
Blood potassium decreased (Investigations) | 0 | 14 | 2 | 8 | 17
Blood sodium increased (Investigations) | 0 | 13 | 10 | 8 | 8
Blood potassium increased (Investigations) | 1 | 16 | 12 | 5 | 2
Lipids increased (Investigations) | 2 | 8 | 3 | 4 | 9
Dyslipidaemia (Metabolism and nutrition disorders) | 5 | 9 | 6 | 10 | 12
Dizziness (Nervous system disorders) | 22 | 28 | 10 | 4 | 3
COVID-19 (Infections and infestations) | 8 | 12 | 6 | 11 | 5
Hyperuricaemia (Investigations) | 2 | 11 | 3 | 5 | 2
Hyperkalaemia (Investigations) | 5 | 8 | 1 | 1 | 2
Dizziness postural (Nervous system disorders) | 7 | 12 | 7 | 6 | 0
Oedema peripheral (General disorders) | 2 | 6 | 4 | 4 | 3
Hypotension (Vascular disorders) | 9 | 0 | 0 | 3 | 0
Hypertension (Vascular disorders) | 3 | 0 | 3 | 1 | 0
Blood triglycerides increased (Investigations) | 2 | 2 | 1 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 2 | 2 | 0 | 0 | 1
Glomerular filtration rate increased (Investigations) | 1 | 0 | 1 | 1 | 0
Blood creatine increased (Investigations) | 1 | 0 | 0 | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 0 | 1 | 0 | 1
Asthenia (General disorders) | 2 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The trial included comparatively few participants with very high levels of blood pressure (BP), which makes direct comparison with previous trials challenging. The trial design did not allow a direct randomized comparison between ½ dose and standard dose combinations, or with other drugs and doses that are in common use. The option of non-uptitration after 6 weeks of half-dose regimens likely led to underestimation of the difference between standard dose regimens.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT04518293/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT04518293/SAP_001.pdf